CLINICAL TRIAL: NCT02287831
Title: Safety and Efficacy of Umbilical Cord Mesenchymal Stem Cell Injection for Peripheral Arterial Disease
Brief Title: Umbilical Cord Mesenchymal Stem Cells Injection for Peripheral Arterial Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Pingping Huang,MD, M.D., Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13ZCZDSY02200
Record Dates: First submitted 2014-11-02; First posted 2014-11-11 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- umbilical cord mesenchymal stem cells (Experimental): Multiple intra muscular injection of mesenchymal stem cells derived from human umbilical cord.
  Interventions: Biological: umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: umbilical cord mesenchymal stem cells

SUMMARY:
The purpose of this study is to assess the safety and efficacy of umbilical cord blood mesenchymal stem cells with peripheral arterial disease.

DETAILED DESCRIPTION:
The present study is designed to implant UCB-MSC in patients with CLI, which are resulted from peripheral arterial disease,such as thromboangiitis obliterans, atherosclerosis obliterans and diabetic foot, and to evaluate the safety and efficacy of the implantation procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-75 years
2. Patients confirmed diagnosed peripheral vascular disease , ankle-brachial index < 0.9
3. Poor distal arterial outflow tract
4. Patient had at least 3 months conservative treatment ,which resulted in little or no improvement
5. Poor physical condition can not tolerate surgery
6. Patients are willing to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Renal function damage (over 2 X upper normal range) Liver function damage (over 3 X upper normal range )
2. Severe or acute organ damage
3. Presence of malignancy
4. Pregnancy or lactating patients
5. HIV positive
6. ABI≧0.9
7. A history of severe allergies related cell therapy
8. Conservative treatment < 3 months
9. Acute limb ischemia
10. Local obvious infection uncontrolled
11. Alcoholics or drug abusers within a year
12. Severe psychiatric disorder.
13. Patients need surgical treatment
14. Above the ankle gangrene
15. Patients with other factors which were considered not to be suitable to participate in the study by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-02; Primary Completion 2022-12 (Actual); Study Completion 2022-12-26 (Actual)

PRIMARY OUTCOMES:
To evaluate safety and tolerability related to the intramuscular injection of autologous Umbilical cord blood derived stem cells. | 6 months
  Amputation rate and mortality will be combined to report safty in %

SECONDARY OUTCOMES:
To evaluate effectiveness related to the intramuscular injection of autologous Umbilical cord blood derived stem cells. | 6 months
  Rest pain, temperature of skin and cold feeling will be combined to report effectiveness in score.

CONTACTS AND LOCATIONS:
Overall Officials: Pingping Huang, M.D., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China